CLINICAL TRIAL: NCT06604637
Title: Effectiveness of Vagus Nerve Stimulation in Individuals With Tension-Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Mesut Arslan, Assistant Professor, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTH-VNS
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Tension-Type Headache
Keywords: Tension-Type Headache; Vagus Nerve Stimulation
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VNS Group (Experimental): In addition to standard treatment, noninvasive transcutaneous auricular vagus nerve stimulation (taVNS) will be applied to this group.
  Interventions: Other: Non-invasive transcutaneous auricular vagus nerve stimulation (taVNS)
- Control roup (No Intervention): The control group will receive standard treatment ( patient education+lifestyle recommendations).

INTERVENTIONS:
Other: Non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) — taVNS will be applied for a total of 12 sessions, 20 minutes each session, 3 days/week.
  Arms: VNS Group

SUMMARY:
It is planned to examine the effect of Vagus Nerve Stimulation on headache symptoms in individuals with tension-type headache.

DETAILED DESCRIPTION:
Tension-type headache is the most common primary headache, usually bilateral, characterized by oppressive and squeezing pain of mild or moderate intensity, unchanged by physical activity. It affects approximately 80% of the population and has a point prevalence of 42% in the general population.

There are various pharmacological and non-pharmacological treatment methods for tension-type headache. One of the non-pharmacological treatment methods may be Vagus Nerve Stimulation (VNS). VNS can affect healing processes by regulating the autonomic nervous system and reduce symptoms in tension-type headache.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with tension-type headache according to the International Classification of Headache Disorders (ICHD-3) criteria,
* Individuals between the ages of 18-65,

Exclusion Criteria:

* History of trauma or surgery to the head and neck region,
* Presence of lesions or metal implants in the application area,
* Uncontrolled hypertension/abnormal ECG results/history of myocardial infarction/pacemaker and similar cardiovascular disease history/suspicion,
* Pregnancy or suspicion,
* Other primary and secondary headache types,
* Individuals who received physiotherapy in the last 6 months,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline at 4 weeks
  In the headache diary, the severity of the pain will be questioned with a numerical pain scale.
Pain duration | Change from baseline at 4 weeks
  The duration of pain will be questioned in the headache diary.
Number of days of pain for 1 month | Change from baseline at 4 weeks
  The number of days of pain during a month will be questioned in the headache diary.
Heart rate variability | Change from baseline at 4 weeks
  Heart rate variability will be measured with an automatic device.

SECONDARY OUTCOMES:
Headache Impact Scale | Change from baseline at 4 weeks
  It is a 6-item scale assessing vitality, pain, psychological state, social, role and cognitive function. The total score of the scale varies between 36-78; higher scores indicate a higher level of impact on the quality of life of the individual.
Depression Anxiety Stress Scale (DASS-21) | Change from baseline at 4 weeks
  It evaluates the condition of the individual in the last week. It is a 21-question questionnaire consisting of 3 subscales: depression, anxiety and stress. The questionnaire score ranges from 0 to 21 for each subgroup. High scores indicate the presence and severity of depression, anxiety and stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren Üniversitesi, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No